CLINICAL TRIAL: NCT00178035
Title: Geriatric Depression: Neurobiology of Treatment
Brief Title: Sleep Deprivation Plus Paroxetine for Treating Major Depression in Elderly Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH037869-02 (NIH); 970356; DATR A4-GPS
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: Depression; Unipolar Depression; Elderly depression; Late-Life
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Paroxetine

INTERVENTIONS:
Drug: paroxetine
Behavioral: One night of Total Sleep Deprivation

SUMMARY:
This study will determine the effectiveness of total sleep deprivation (TSD) for one night plus paroxetine versus either TSD plus placebo or paroxetine alone in inducing rapid symptom resolution of major depression in the elderly.

DETAILED DESCRIPTION:
The clinical response to antidepressant treatment in the elderly is variable and often slow, and difficult to predict reliably before 4-5 weeks of treatment. The delayed onset of antidepressant activity is particularly problematic in the elderly, prolonging the duration of suffering and disability, reducing compliance, and increasing the risk for attempted and completed suicide.

This study seeks to develop a method for effective rapid treatment of major depressive episodes in the elderly and to improve early identification of treatment non-responders, by combining sleep deprivation (for one night) and paroxetine as probes of treatment response and treatment resistance.

This is an experimental study that is randomized, double-blind, and placebo-controlled. We will recruit 158 elderly depressed patients with current major depressive episodes and randomly assign 36 patients to each of three interventions: 1)TSD + paroxetine; 2)TSD + placebo; and 3)paroxetine alone without TSD). The duration of the experimental phase of the study is 17 days: 3 days for pre-treatment sleep studies and 14 days for initial paroxetine or placebo treatment under double-blind conditions.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00177294

http://clinicaltrials.gov/show/NCT00178074

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Current episode of unipolar, major depression
* HRSD (17 item)score of 15 or higher
* Folstein Mini-Mental Status exam score of 17 or higher

Exclusion Criteria:

* Lifetime diagnosis of any psychotic disorder
* Lifetime diagnosis of bipolar disorder

  _Alcohol or drug abuse within the past 6 months
* Contraindication to treatment with SSRI therapy
* History of seizure disorder
* Baseline apnea/hypopnea index of 20 or higher
* Hyponatremia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158
Dates: Start 1999-12; Study Completion 2003-08

PRIMARY OUTCOMES:
Combined treatment of total sleep deprivation(TSD)for one night + paroxetine will be superior to the combination of placebo + TSD and to paroxetine alone (without TSD)in bringing about rapid resolution of depressive symptoms.

SECONDARY OUTCOMES:
EEG Sleep measures
Cognitive status: Folstein Mini-Mental Status Exam, and CDR
Quality of Life measures: Quality of Wellbeing Scale, CIDI Health Services Utilization, OARS, GAF, PSQI, SF-36, UKU, and CIRS-G
Social Support: Interpersonal Support Evaluation List, Luben Social Network Scale
Psychiatric status: SCID, Hamilton Depression Rating Scale, Suicidal History Questionnaire, Antidepressant Treatment History Form, Brief Psychiatric Rating Scale, and anxiety subscale of Brief Symptom Inventory
MRI

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Reynolds III, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States